CLINICAL TRIAL: NCT03733028
Title: Developing a Mobile Intervention for Veterans With PTSD and Problematic Anger
Brief Title: Mobile Intervention for Veterans With PTSD and Anger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2965-W
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Posttraumatic Stress Disorder; Anger
Keywords: anger; posttraumatic stress disorder; hostile interpretation bias; mHealth
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobile Intervention for Reducing Anger (MIRA) (Experimental): Participants in this arm will be provided with a device that has the MIRA application (app) and asked to use the app for a period of 4 weeks.
  Interventions: Behavioral: Mobile Intervention for Reducing Anger (MIRA)
- Mindfulness Intervention (Active Comparator): Participants in this arm will be provided with a device that has the Mindfulness application (app) and asked to use the app for a period of 4 weeks.
  Interventions: Behavioral: Mindfulness Intervention

INTERVENTIONS:
Behavioral: Mobile Intervention for Reducing Anger (MIRA) — This is a mobile intervention that uses interpretation bias modification (IBM) techniques to reduce the hostile interpretation bias. Participants will be given a mobile device with the MIRA app and instructed to complete 5 treatment sessions each week for a period of 4 weeks. Each session takes approximately 10 minutes. The app also includes a Nightly Diary to track symptoms, a calendar to program session reminders, and a My Progress feature to track use and performance.
  Arms: Mobile Intervention for Reducing Anger (MIRA)
Behavioral: Mindfulness Intervention — This is a mobile intervention that uses the Mindful Breathing and Body Scan exercises from the "Mindfulness Coach" app. These audio-guided exercises take approximately 10 minutes each. Participants will be given a mobile device with the Mindfulness app and instructed to complete 5 exercises (i.e., Body Scan or Mindful Breathing) each week for a period of 4 weeks. The app also includes a Nightly Diary to track symptoms, a calendar to program reminders, and a My Progress feature to track use and performance.
  Arms: Mindfulness Intervention

SUMMARY:
Anger is the mostly commonly reported reintegration concern among combat Veterans, especially those with PTSD. Problematic anger is associated with significant functional impairment. In the current project, the investigators will pilot-test a newly developed mobile app, entitled Mobile Intervention for Reducing Anger (MIRA), among Veterans with PTSD and problematic anger. The project will compare the MIRA app to a contact control condition. The investigators hypothesize that Veterans with PTSD and problematic anger will find the MIRA app acceptable and will be willing to use it to reduce their anger difficulties and improve psychosocial and occupational functioning.

DETAILED DESCRIPTION:
Anger is the mostly commonly reported reintegration concern among combat Veterans, especially those with PTSD. Problematic anger is associated with significant functional impairment. One of the mechanisms associated with problematic anger and aggression is hostile interpretation bias, i.e., a tendency to interpret ambiguous interpersonal situations as hostile. The investigator has previously developed and piloted a computer-based interpretation bias modification intervention that successfully reduces both hostile interpretation bias and anger outcomes. In the current project, the investigators will pilot-test a mobile application version of the existing computer-based intervention, entitled Mobile Intervention for Reducing Anger (MIRA), among Veterans with PTSD and problematic anger. The project will compare the MIRA app to a contact control condition to evaluate the feasibility of recruitment, randomization, and retention procedures. The investigators will also utilize psychophysiological and electronic diary monitoring to determine whether this assessment could be used as an outcome or mechanistic variable in a subsequent randomized clinical trial application focused on evaluating the efficacy of the MIRA intervention.

ELIGIBILITY:
Inclusion Criteria:

* Veterans diagnosed with PTSD, established via the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5)
* Reporting a score of 12 on the 5-item Dimensions of Anger Reactions Scale
* Able to read at least 6th grade level material

Exclusion Criteria:

* Expect to be unstable on their medication regimen during the study
* Currently in a period of active psychosis or mania
* Exhibit current prominent suicidal or homicidal ideation requiring immediate intervention
* Receiving (or plan to receive) other anger management psychotherapy or trauma-focused therapy for PTSD (i.e., prolonged exposure, cognitive processing therapy during the course of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten H Dillon, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mobile Intervention for Reducing Anger (MIRA) | Mindfulness Intervention
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Intervention for Reducing Anger (MIRA) | Mindfulness Intervention | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.56 (12.82) | 59.29 (10.76) | 54.53 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 14 | 11 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 7 | 19
  White | 2 | 5 | 7
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Measured by Percentage of Recruitment Goal Met
Description: Patient recruitment goal feasibility goal will be met if recruitment is 75% or greater of recruitment expectation. Recruitment expectation is 20 in each arm.
Time Frame: Through study completion (approximately 2 years)
Population: 20 participants per arm was the expected number of participants to be recruited.
Measure: Number; unit: participants
Arm/Group | Mobile Intervention for Reducing Anger (MIRA) | Mindfulness Intervention
Number analyzed (Participants) | 20 | 20
participants | 16 | 14

2. Primary Outcome: Number of Participants Lost to Attrition During Treatment
Description: Treatment retention feasibility goal will be met if attrition from MIRA treatment arm is no more than 25%.
Time Frame: Post-treatment assessment visit (approximately one month after enrollment)
Population: This population is defined as all participants who began treatment.
Measure: Number; unit: participants
Arm/Group | Mobile Intervention for Reducing Anger (MIRA) | Mindfulness Intervention
Number analyzed (Participants) | 16 | 14
participants | 0 | 1

3. Primary Outcome: Number of Participants Who Report Satisfaction With the MIRA App
Description: Patient satisfaction goal will be met if 80% or greater of participants indicate that they are either "very satisfied" or "mostly satisfied" with the MIRA app on item #7 of the Client Satisfaction Questionnaire.
Time Frame: Post-treatment assessment visit (approximately one month after enrollment)
Population: These are all participants assigned to the MIRA group who completed treatment.
Measure: Number; unit: participants
Groups:
- MIRA Group/Users Only: This outcome only applies to participants in the MIRA group, as they were the only ones to use the MIRA app.
Arm/Group | MIRA Group/Users Only
Number analyzed (Participants) | 16
participants | 14

4. Primary Outcome: Average Number of Treatment Sessions Completed by MIRA App Users
Description: Our App utilization goal will be met if MIRA app utilization rates are greater than 50% of expected use. Expected use is defined as 20 sessions completed, and the app utilization goal will be met if participants complete, on average, at least 10 sessions.
Time Frame: Post-treatment assessment visit (approximately one month after enrollment)
Population: These are all participants assigned to the MIRA group who completed treatment. One participant was withdrawn prior to beginning treatment, and another withdrew during treatment.
Measure: Mean (Standard Deviation); unit: sessions completed
Arm/Group | MIRA Group/Users Only
Number analyzed (Participants) | 16
sessions completed | 17.13 (8.79)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for approximately 17 weeks, from baseline to the 3-month follow-up visit.
Arm/Group | Mobile Intervention for Reducing Anger (MIRA) | Mindfulness Intervention
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 2/16 | 4/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mobile Intervention for Reducing Anger (MIRA) (N=16) | Mindfulness Intervention (N=14)
Distress upon completing interview about posttraumatic stress disorder symptoms (Psychiatric disorders) | 1 (1) | 1 (1)
frustration/discomfort with using the mobile app (General disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT03733028/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT03733028/ICF_001.pdf